CLINICAL TRIAL: NCT02087787
Title: Establishing a BMT Legal Clinic to Support Patients With Cancer Undergoing Blood or Marrow Transplant
Brief Title: Medical-legal Partnership (MLP) to Support Bone Marrow Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013NTLS112
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Blood or Marrow Transplant
Keywords: bone marrow transplant; hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will be provided the standard method, which is providing the Cancer Legal Line (CALL) brochure with a short explanation of the resource.
- Intervention (Experimental): The intervention group will be provided with a 2 hour consultation with an attorney in the BMT Legal Clinic with potential follow-up as needed.
  Interventions: Behavioral: BMT Legal Clinic

INTERVENTIONS:
Behavioral: BMT Legal Clinic — 2 hour consultation with an attorney in the BMT Legal Clinic with potential follow-up as needed.
  Arms: Intervention

SUMMARY:
The goal of this study is to develop and test the effects of a marrow transplant (BMT) Legal Clinic established through a medical-legal partnership (MLP) in an adult blood and marrow (BMT) transplant setting. This will be a 2-arm randomized, controlled clinical trial, in which the intervention group of patients will participate in a BMT Legal Clinic and the control group is provided standard information regarding legal resources.

DETAILED DESCRIPTION:
Blood or marrow transplant patients (BMT) may experience legal support needs through their transplant process. Specific examples of medical-legal issues impacting BMT patients include social security disability benefits, Will/estate issues, employment concerns, and creditor issues. At the beginning of the transplant process, BMT patient-families are often overwhelmed by the stress of transplant, and their focus is usually on their care and treatment needs. Legal planning that may be important to patient-families may not be considered or deferred.

Presently, the process of referral to legal services is predominantly a reactive process. Once a patient identifies a legal issue or concern to a BMT social worker, this is often after the issue escalates to the point where it creates significant stress for the patient-family. The BMT social workers have prolonged contact with these patients and frequently spend many hours trying to assist patients to resolve these issues.

Cancer Legal Line (CALL) provides caring and compassionate pro bono legal consultation and other referral or pro-bono legal services based on income guidelines to Minnesotans affected by cancer. CALL has provided this support based on Blood and Marrow Transplant (BMT) social work referral for the past 5 years. To our knowledge, there have been no medical-legal partnerships established within hospitals for patients undergoing blood or marrow transplant with cancer.

It is hypothesized that by establishing an onsite BMT Legal Clinic through a Medical-Legal Partnership (MLP), that patient-and families can be better served through proactive legal consultation. The BMT Legal Clinic would serve to connect the CALL staff with the BMT care team to better serve patients to address patients' concerns, promote well-being, and reduce stress related to medical-legal issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old, who have been identified by the BMT social worker as having a cancer or pre-cancer diagnosis and are Minnesota residents with potential legal needs (see the list below), expected to proceed to transplant, considered the primary client for legal services or are at least 18 years old and have a legal-designate.
* The patient or legal designate must be able to complete study tools by the BMT social workers. Interpreters will be provided by UMMC for non-English speaking pt's and BMT social workers will assist patients who cannot read.
* Patients must have interest in a legal consultation as specified by the I-Help model to receive free legal consultation.

Exclusion Criteria:

* Patients who do not have any identified any potential legal needs, or whose legal needs are beyond those covered in the I-Help model.
* Patients with non-cancer diagnoses, as CALL only provides services for cancer or pre-cancer diagnoses.
* Patients who are not residents of Minnesota as CALL attorneys are only licensed to practice law in Minnesota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Difference between Concern and Well-being score | 100 days
  The difference between the Concern and Well-being score from baseline to post-transplant (MyCaW scale)

SECONDARY OUTCOMES:
Proportion of patients with specific legal concerns | 100 days
  Proportion of patients with specific legal concerns
Mean cost of legal services | 100 days
  Cost of legal services over 100 days post transplant
Proportion of patients satisfied | 100 days
  Self-reported assessment of patient satisfaction using the proportion of patients who were satisfied or very satisfied with the legal services by day 100 post transplant
Average PSS-10 score | 100 days
  Average score on PSS-10 stress scale
Number of hours on legal service | 100 days
  Number of hours spent on legal service for 100 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Parran, MS, RN, Principal Investigator — University of Minnesota Medical Center, Fairview
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States